CLINICAL TRIAL: NCT04346940
Title: The Effectiveness of Telerehabilitation-Based Exercises in Elderly People Under Social Isolation Process Due to Coronavirus
Brief Title: The Effectiveness of Telerehabilitation-Based Exercises in Elderly People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Telerehabilitation; Elderly People; Social Isolation
Keywords: COVID-19; Exercise
MeSH Terms: conditions — Social Isolation; COVID-19; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The group to which the exercise protocol consisting of chair-based exercises will be applied.
  Interventions: Other: Telerehabilitation
- Control Group (Active Comparator): Group to be given an exercise brochure
  Interventions: Other: Exercise brochure

INTERVENTIONS:
Other: Telerehabilitation — 15 volunteers aged 65 and over will be included in this group. An online exercise program has been created for individuals who will participate in the study. It is planned that this program will continue for 3 days a week, 6 weeks, and the duration of exercise will reach 45 minutes in the last week due to the increase in the number of repetitions about 30 minutes at the beginning. The treatment sessions will start with warm-up exercises, complete with posture exercises, joint range of motion exercises, stretching exercises, and cool-down exercises in the main program.
  Arms: Study Group
Other: Exercise brochure — The same exercises will be given to the control group as a brochure and they will be asked to do it for 6 weeks.
  Arms: Control Group

SUMMARY:
An epidemic of pneumonia , which is thought to have developed due to a new coronavirus, was detected in Wuhan, Hubei Province of the People's Republic of China, and this epidemic could not be brought under control, leading to other provinces of China in a short time and then to a pandemic. It has spread all over the world including the European continent. Causative Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) and the disease caused by the new virus (novel) coronavirus-2019 (2019-nCoV) and subsequently the COVID-19. After the virus was officially detected in our country on 11 March 2020, the number of cases increased rapidly and the virus was isolated in 670 patients within 10 days. The group that is most affected by the outbreak and has the highest mortality rate is the elderly with known cardiovascular diseases. It is important to ensure the social isolation of elderly patients and to minimize all hospital applications as much as possible if they do not have life-threatening urgent problems. To this end, Turkey on 21 March 2020, 65 years of age and older people and patients with chronic curfew was implemented.

Individuals moving away from social life are dealing with their body more, their level of depression and anxiety increase, and their physical functions decrease. The therapy service is offered to people who cannot travel with telerehabilitation, which is defined as the transmission of rehabilitation service to long distances by using electronic information and communication technology.

The purpose of this study is to investigate the effects of telerehabilitation exercises given to elderly individuals on sleep quality, quality of life and balance within the scope of geriatric rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over,Mini Mental Status Scale 24 and above, To be able to communicate verbally and visually,Those who do not have serious heart disease (aortic stenosis, angina, hypertrophic cardiac myopathy, arrhythmia, pacemaker) that may prevent exercise,Having the necessary technological competence to provide remote video communication at home,To be at least 20 m ambassador

Exclusion Criteria:

* Mini Mental Status Scale being lower than 24,Those with serious heart disease (aortic stenosis, angina, hypertrophic cardiac myopathy, arrhythmia, pacemaker) that may interfere with exercise,Visual or auditory loss

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-10 (Estimated); Primary Completion 2020-10-10 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Standardized Mini Mental Test | 2 weeks
  Screening test in which cognitive functions are evaluated globally. With standardized mini mental test, the patient is evaluated under 5 main topics. The patient receives a maximum of 30 minimum 0 points at the end of the test. The critical score here is 27 or 24. It is decided that patients scoring below 24 have cognitive impairment. In some cases, the limit is considered to be 27 points.
Mini Nutritional Assesment | 2 weeks
  The Mini Nutritional Assessment (MNA) has recently been designed and validated to provide a single, rapid assessment of nutritional status in elderly patients in outpatient clinics, hospitals, and nursing homes. sum of the MNA score distinguishes between elderly patients with: 1) adequate nutritional status, MNA ≥ 24; 2) protein-calorie malnutrition, MNA < 17; 3) at risk of malnutrition, MNA between 17 and 23.5.
Short Physical Performance Test | 2 weeks
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Single Leg Stance Test | 2 weeks
  The one-leg standing (OLS) test is one of the balance tests used to diagnose musculoskeletal ambulation disability symptom complex (MARS), a condition newly defined by three professional Japanese medical societies in 2006 to help identify the symptoms of motor organ deterioration and establish preventive strategies. Although many studies have used the OLS test, none has shown conclusively that the test can be used as a practical marker of frailty among elderly people, especially in community settings.
Charlson Comorbidity Index | 2 weeks
  Scaling that can be applied with the informer or by obtaining information from the medical records in order to quantify the comorbidities and to examine their effects on prognosis in clinical studies. 19 disease states are evaluated.
Clinic Fragility Scale | 2 weeks
  A multi-dimensional loss of reserve that leads to fragility, fragility (energy, physical ability, cognition,health) syndrome and weakness 3 or more symptoms (unintentional weight loss, feeling tired, weak grip, slow walking rate and low physical activity), the person can be described as we It consists of 9 questions.If there are 3 or more symptoms (unintentional weight loss, fatigue, poor grip, slow walking speed, and low physical activity), the person can be described as weak.
Pittsburgh Sleep Quality Index | 2 weeks
  It is a scale evaluating sleep quality with a total of 19 questions under 7 main topics. Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report scale that evaluates sleep quality and disorder in the past month The total score of the 7 components gives the scale total score. The total score ranges from 0-21. A total score greater than 5 indicates "poor sleep quality".
Social Isolation Survey | 2 weeks
  Social participation levels were evaluated with the Social Isolation Survey. Minimum 0 and maximum 24 points are obtained from the scale. 0 points indicate complete social isolation while 24 points indicate high social relationship. A value of 0-10 indicates complete social isolation, 12-15 isolation, 16-18 partial isolation, 19-21 social, 21-24 high social relationship Quality of life scale in the elderly
Quality of life scale in the elderly | 2 weeks
  The Quality of life scale in the elderly (CASP-19) was developed in 2003 to measure.The scale consists of 19 items and "Control", "Autonomy", "Pleasure" and "Self-realization." Each item of the original scale is "never" (0 score) to "always" (3 points) It is rated as a 4-point Likert type. The increase in the total score indicates that the quality of life increases.
The Physical Activity Scale for the Elderly | 2 weeks
  Physical Activity Scale for the Elderly (PASE) is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiological studies of persons age 65 years and older. The overall PASE score ranges from 0 to 400 or more and high scores show better physical activity levels.
Timed Up and Go Test | 2 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require
30 Second Chair Stand Test | 2 weeks
  The 30-s Chair Stand Test (CST) consists of standing up and sitting down from a chair as many times as possible within 30 seconds. A standard chair without backrest, but with armrests is used. Initially, the person is seated on the chair with his backs upright. They are told to look forward with their arms folded in their chest and rise at their preferred speed after the command "1, 2, 3, go". All trials must be carried out using the same chair and similar environmental conditions.
The Beck Depression Inventory | 2 weeks
  The Beck Depression Inventory (BDI) is a 21-item, self-rated scale that evaluates key symptoms of depression. Individual scale items are scored on a 4-point continuum (0=least, 3=most), with a total summed score range of 0-63. Higher scores indicate greater depressive severity. Two subscales include a cognitive-affective subscale and a somatic-performance subscale.
The Beck Anxiety Inventory | 2 weeks
  The Beck Anxiety Inventory (BAI) is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults.The questions used in this measure ask about common symptoms of anxiety . It is designed for individuals who are of 17 years of age or older and takes 5 to 10 minutes to complete. Several studies have found the Beck Anxiety Inventory to be an accurate measure of anxiety symptoms in children and adults.

IPD SHARING:
Plan to Share IPD: No